CLINICAL TRIAL: NCT05715450
Title: Falciformopexy for Treatment Perforated Peptic
Brief Title: Falciformopexy for Treatment Perforated Peptic Ulcer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Hamada, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Falciform ligament on PPU
Record Dates: First submitted 2022-09-29; First posted 2023-02-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Perforated Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Falciformopexy for Treatment Perforated Peptic Ulcer (Other): Use falciform ligament flap for repair perforated peptic ulcer
  Interventions: Procedure: Falciformopexy for Treatment Perforated Peptic Ulcer

INTERVENTIONS:
Procedure: Falciformopexy for Treatment Perforated Peptic Ulcer — use the falciform ligament on perforated peptic ulcer

SUMMARY:
Use the falciform ligament flap for the treatment of perforated peptic ulcer

DETAILED DESCRIPTION:
Peptic ulcer perforation (PUP) is one in all the foremost common critical surgical emergencies. The omentum flap is usually wont to cover a PUP. However, the omentum can not be utilized in cases of severe peritonitis or previous surgical removal. this is often the primary study conducted in Vietnam that was designed to analyse the outcomes of patients with PUPs who were treated using the ligament.

In the population, the prevalence of ulcer disease supported physician diagnosis ranges from 0.12% to 1.50%, and hospitalization rates range from 0.10% to 0.19%. ulceration perforation (PUP) is one of the foremost common surgical emergencies worldwide, which is necessitate emergent surgical intervention.

the death rate of PUPs is between 1.3% and 20%, and mortality thanks to a perforation of a gastric ulcer is over mortality because of a perforation of a duodenal ulcer (40% vs 10%) . Some studies have shown that having comorbidities, being over 70 years old, undergoing surgical procedure after 36 h, PUP diameter greater than 1 cm2 and postoperative com- plications are associated with mortality. The technique of using the omental patch for repair PUP is commonest now thanks to mobility and vascularity but is also using the falciform ligament in some cases due to highly vascularity.

The technique of using the falciform ligament for the treatment of PUPs was reported in 1978 by Fry . The purpose of the study was to explain the technique and therefore the results of using the falciform ligament for the treat- ment of PUPs during a large volume surgical centre in Assuit university hospital found the falciform patch to be a successful technique in repair PUP and is assumed to be as effective as omental patch but more advantage because of highly vascular.

ELIGIBILITY:
Inclusion Criteria:

- Any cases presented with PPU within age from 18 till 70 years.

Exclusion Criteria:

* malignancy.
* Previous GIT and liver surgery.
* nonoperative treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Falciformopexy for Treatment Perforated Peptic Ulcer | Baseline
  The aim is to decrease incidence of leakage from the perforated peptic ulcer by using the falciform ligament for repair of the perforated peptic ulcer.
  Firstly, the investigator will seek to repair the perforation using suture to approximate edges then use falciform ligament as a secound layer to ensure security and prevent postoperative leakage that will lead to peritonitis and death.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Hamada Abd elbaset, Principal Investigator — Assiut University

REFERENCES:
- [Background] Fry DE, Richardson JD, Flint LM Jr. Closure of an acute perforated peptic ulcer with the falciform ligament. Arch Surg. 1978 Oct;113(10):1209-10. doi: 10.1001/archsurg.1978.01370220095016. PMID 708243
- [Background] Son TQ, Hoc TH, Huong TT, Long VD, Tung TT, Quyet NC, Panha L, Van Chi N. Outcomes of surgical management of peptic ulcer perforation using the falciform ligament: A cross-sectional study at a single centre in Vietnam. Ann Med Surg (Lond). 2021 Jun 16;67:102477. doi: 10.1016/j.amsu.2021.102477. eCollection 2021 Jul. PMID 34188907
- [Background] Sung JJ, Kuipers EJ, El-Serag HB. Systematic review: the global incidence and prevalence of peptic ulcer disease. Aliment Pharmacol Ther. 2009 May 1;29(9):938-46. doi: 10.1111/j.1365-2036.2009.03960.x. PMID 19220208